CLINICAL TRIAL: NCT02368613
Title: A Clinical Trial for Evaluation of Adequate Dose and Safety of DW-3102 in Hypercholesterolemia Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW-3102_201
Record Dates: First submitted 2015-02-15; First posted 2015-02-23 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- placebo group (Placebo Comparator): Placebo
  Interventions: Drug: DW-3102
- test1 group (Active Comparator): DW-3102 125mg
  Interventions: Drug: DW-3102
- test2 group (Active Comparator): DW-3102 250mg
  Interventions: Drug: DW-3102
- test3 group (Active Comparator): DW-3102 500mg
  Interventions: Drug: DW-3102

INTERVENTIONS:
Drug: DW-3102

SUMMARY:
The purpose of this study is to evaluate adequate-dose of DW-3102 in the treatment of hypercholesterolemia patients by conducting phase 2a. 4 groups involving placebo group, each groups are composed by 16, will be participated in this trial.

ELIGIBILITY:
Inclusion Criteria:

* More than 19 years old
* Those who meet the fasting serum lipid levels along table
* Those who are under 350 mg/dL of TG level when fasting

Exclusion Criteria:

* The patient of acute arterial disease
* The patient of severe heart failure(NYHA class III or IV)
* Within the last 6 months clinically meaningful treatment that requires that arrhythmias or cardiac conduction disorders
* Uncontrolled hypertension ( systolic blood pressure ≥ 180mmHg or diastolic blood pressure ≥ 110mmHg or more later)
* Endocrine or metabolic disease patients known to affect serum lipids or lipoproteins
* Fibromyalgia, myopathy, rhabdomyolysis, or sudden muscle pain or have in the past, such as statin (HMG CoA reductase inhibitors) in patients with muscle -related adverse drug experience of the system
* Drug malabsorption by gastrointestinal surgery experience (but simple appendectomy and hernia surgery is excluded) or gastrointestinal disorders ( Crohn's disease , ulcers , acute or chronic pancreatitis , etc. )
* Patients with history of malignancies including leukemia and lymphoma within the past five years
* If severe renal impairment or in patients with impaired liver and hematological findings following the same
* Patients who have participated in another clinical trial within the previous 30 days or Prior to the administration of at least five times the half-life of the active ingredient is not elapsed patient IND
* Those having a known hypersensitivity to hyperlipidemia treatment
* Patients with hypersensitivity or allergy to cruciferous plants
* Patients with a history of drug or alcohol abuse within the last 12 months
* Female patients of childbearing age
* In the case of male test subjects , if the spouse does not agree with the use of childbearing age when women work , recognized contraception exclusion criteria presented in Section 15
* Patient who are inappropriate by investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
The change of LDL-C% | 6 weeks